CLINICAL TRIAL: NCT05386771
Title: The Effect of Ingesting a Whey and Collagen Protein Blend on Myofibrillar and Connective Tissue Protein Synthesis Rates at Rest and During Recovery From Exercise
Brief Title: Effects of Whey and Collagen Protein Blend on Protein Synthesis Rates
Acronym: Blend
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: METC 22-017
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2022-09

CONDITIONS: Muscle Protein Synthesis
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Double-blind, parallel-group, placebo-controlled intervention study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomized double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whey and collagen protein blend (Experimental): A blend of 25g of whey protein and 5g of collagen protein
  Interventions: Dietary Supplement: Whey/collagen protein blend; Behavioral: Resistance exercise
- Placebo (Placebo Comparator): Water, same volume as the experimental study beverage
  Interventions: Dietary Supplement: Whey/collagen protein blend; Behavioral: Resistance exercise

INTERVENTIONS:
Dietary Supplement: Whey/collagen protein blend — Ingestion of 30g of protein dissolved in 300ml water consumed after an exercise session
Behavioral: Resistance exercise — A single resistance exercise session of the leg press and leg extension exercise

SUMMARY:
Rationale: Protein ingestion stimulates muscle protein synthesis and augments the muscle protein synthetic response to a single exercise session. In support, protein supplementation has been shown to augment the gains in muscle mass and strength following resistance exercise training. The force generated by contracting muscle is transferred through a network of connective tissue proteins towards the bone. Consequently, remodeling of skeletal muscle connective tissue represents an essential component of skeletal muscle adaptation to exercise. The anabolic effect of a protein supplement is mainly determined by the plasma amino acid response after ingestion. Although whey protein is considered the preferred protein source to maximize myofibrillar protein synthesis rates, it contains insufficient glycine and proline to support the post-exercise increase in connective tissue protein synthesis rates. In contrast, collagen protein is rich in glycine and proline and has, therefore, been proposed as a preferred protein source to support connective tissue remodeling. Hence, the combined ingestion of whey plus collagen protein may therefore be preferred to stimulate both myofibrillar and collagen protein synthesis rates in skeletal muscle tissue. The most ideal protein supplement for stimulating both myofibrillar and collagen protein synthesis is one that gives a rapid initial rise in plasma amino acid concentrations including leucine, proline and glycine concentrations. However, the effect a blend of whey and collagen protein on myofibrillar and connective tissue protein synthesis rates is unknown.

Objective: To assess the effect of a whey and collagen protein blend versus a placebo on myofibrillar and connective tissue protein synthesis rates in muscle obtained during recovery from exercise and rest in vivo in humans.

Study design: Double-blind, parallel-group, placebo-controlled intervention study.

Study population: 28 healthy recreationally active males (18-35 y; BMI: 18.5-30 kg/m2).

Intervention: Participants will perform unilateral resistance exercise followed by the ingestion of either a blend of 25 g whey and 5 g collagen protein or a non-caloric placebo (flavored water). Continuous intravenous stable isotope amino acid tracer infusions will be applied, and plasma and muscle samples will be collected in order to assess protein synthesis rates in muscle tissue.

DETAILED DESCRIPTION:
This study utilizes a double-blind, parallel-group, placebo-controlled intervention with two groups. In total, up to 38 healthy recreationally active male subjects (age: 18-35 y) will be included in the study, while 28 subjects need to finish the experimental test day. Subjects will perform a single unilateral resistance exercise session (leg press and leg extension) and will be randomly assigned to consume a beverage containing either a blend of 25 g whey and 5 g collagen protein or a placebo with non-nitrogenous, non-caloric flavored water. Blood and muscle biopsies will be collected while a primed continuous infusion of L-[ring-13C6] phenylalanine infusion will be administered. The duration of the entire study will be approximately 24 months. This period includes screening, testing and data analysis of all 28 subjects. Subject testing will be done after approximately 12 months.

Subjects will participate in one screening session. During this session, the study procedures will be explained again verbally and any remaining questions by the subject will be answered. Thereafter, the informed consent form will be signed. Subjects will be asked to fill in a medical questionnaire to gather information about their general health, medical history, use of medication and sports activities. Body height , body weight and body composition will be measured. The BIA is a simple and non-invasive procedure. Finally, subjects will be familiarized and tested for strength on the exercise machines (leg-press and leg-extension). Subjects will be instructed on proper single legged weight-lifting technique on each exercise machine (leg-press and leg-extension) and complete a standardized testing protocol to determine a measurement of maximal strength (1RM) on each exercise machine. The testing protocol requires that the subjects complete sets on each exercise machine increasing in weight until volitional fatigue occurs. The heaviest weight that could have been lifted with good execution of the exercise will be taken as the 1RM. Following the determination of 1RM, subjects will be scheduled for their experimental testing day.

All subjects will consume a standardized dinner the evening before each test day. The subjects will receive the meal after the screening test in a thermal bag. The subjects will be instructed to store the meal in a freezer until preparation and to prepare the meal themselves according to the instructions on the label. All subjects will be instructed to refrain from any sort of heavy physical exercise and alcohol intake 2 days before the test day. In addition, subjects will be asked to record their food intake and physical activity for 48 h before the start of the test day in a diary that will be provided during the screening.

Each subject will participate only in 1 experimental test day, which lasts ~9 h. The protocol is designed to assess the post-exercise plasma amino acid responses, myofibrillar and connective tissue protein synthesis.

A general overview of the study protocol is shown in Figure 1. At 7:45 am, following an overnight fast, subjects will arrive at the laboratory by car or public transportation. Subjects will rest in a supine position and a Teflon catheter will be inserted in a heated dorsal hand vein and placed in a hot-box (60°C) for arterialized blood sampling. In the contralateral arm, another Teflon catheter will be inserted for stable isotope infusion. A basal arterialized venous blood sample will be collected (t = -210 min), after which a single intravenous dose of L-[ring-13C6] phenylalanine (Cambridge Isotopes, Andover, MA) will be administered. Thereafter, a continuous infusion of L-[ring-13C6] phenylalanine will be started (t = -210 min) using a calibrated space plus infusomat pump (Braun, Melsungen, Germany), running for 510 min. A muscle biopsy from the upper leg that will not perform the unilateral exercise session will be collected at t = -180 min as a reference to assess post-absorptive muscle protein synthesis rates. After the first muscle biopsy was performed, muscle thickness of the rectus femoris muscle will be measured via ultrasound. Arterialized venous blood samples will be collected at t = -210, -180, -120, -60 and 0 min. At t = -45 min, a unilateral exercise, that consists of 4 sets of 8 repetitions on the leg press and leg extension machine at 80% 1RM 8 reps and last set until failure, will be performed. At t = 0 min muscle biopsies will be collected from the vastus lateralis muscle of both the rested and exercised leg. Immediately following blood collection (t = 0 min), subjects will ingest a test drink containing a blend of 25 g whey and 5 g collagen protein (PRO) or a non-caloric placebo (CON). Following ingestion of the test drink, arterialized venous blood samples will be collected at t = 30, 60, 90, 120, 180, 240 and 300 min. Furthermore, an additional muscle sample will be collected from the rested and exercised leg at t = 300 min.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Aged between 18-35 years
* Healthy, recreationally active (performing exercise 3 times per week or less in the past 6 months)
* BMI 18.5 - 30 kg/m2
* No physical limitations (i.e. able to perform all activities associated with daily living in an independent manner).

Exclusion Criteria:

* Females
* Musculoskeletal disorders
* Use of any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescribed acne medications).
* Participation in any structured regular exercise program
* Chronic use of gastric acid suppressing medication or anti-coagulants
* Pathologies of the gastrointestinal tract
* Blood donation in the past 2 months

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis rates exercised leg | 0-5 hours
  Muscle protein synthesis rates are calculated using L-ring-13C6-phenylalanine tracer and provided as 1 integrated value over the specified timeframe using plasma as precursor of the exercised leg.
Muscle protein synthesis rates rested leg | 0-5 hours
  Muscle protein synthesis rates are calculated using L-ring-13C6-phenylalanine tracer and provided as 1 integrated value over the specified timeframe using plasma as precursor of the rested leg.

SECONDARY OUTCOMES:
Muscle protein synthesis rates | -3-0 hours
  Muscle protein synthesis rates are calculated using L-ring-13C6-phenylalanine tracer and provided as 1 integrated value over the specified timeframe using plasma as precursor.
Plasma glucose concentrations | 0-5 hours
  Plasma glucose concentrations
Plasma insulin concentrations | 0-5 hours
  Plasma insulin concentrations
Plasma amino acids concentrations | 0-5 hours
  Plasma amino acids concentrations

OTHER OUTCOMES:
Age | baseline
  Age in year
Dietary macronutrient intake | 2 days before test days
  assessed by written dietary intake records
Body mass in kg | baseline
  Scale
height in m | baseline
  stadiometer
BMI in kg/m^2 | baseline
  calculated form height and body mass
Whole body lean mass in kg | baseline
  BIA
bodyfat% | baseline
  BIA
1RM | baseline
  maximum strength of both legs

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Centre+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aussieker T, Kaiser J, Hermans WJH, Hendriks FK, Holwerda AM, Senden JM, VAN Kranenburg JMX, Goessens JPB, Braun U, Baar K, Snijders T, VAN Loon LJC. Ingestion of a Whey Plus Collagen Protein Blend Increases Myofibrillar and Muscle Connective Protein Synthesis Rates. Med Sci Sports Exerc. 2025 Mar 1;57(3):544-554. doi: 10.1249/MSS.0000000000003596. Epub 2024 Nov 6. PMID 39501478